CLINICAL TRIAL: NCT05073627
Title: The Effect of Dicloxacillin on Oral Absorption of Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AKF-400; 2021-003814-37 (EudraCT Number)
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers; Drug-drug Interaction
Keywords: P-gp transporter, Induction of P-gp transporter
MeSH Terms: interventions — Dicloxacillin; Dabigatran

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): The investigators measure the baseline of dicloxacillin and the probe drug dabigatran etexilate.
- Dicloxacillin treatment (Experimental): The investigators measure the concentration of dicloxacillin after 9 and 27 days and the concentration of dabigatran after 10 and 28 days of continuously taking dicloxacillin.
  Interventions: Drug: Dicloxacillin

INTERVENTIONS:
Drug: Dicloxacillin — Healthy volunteers will take 2x500 mg dicloxacillin 3 times a day for 30 days. The investigators will measure the baseline concentration of dabigatran and dicloxacillin before start of 30 days of dicloxacillin treatment. On day 9 and 27 the investigators will measure the concentration of dicloxacillin. On day 10 and 28 the investigators will measure the concentration of dabigatran.
  Other Names: Dabigatran etexilate
  Arms: Dicloxacillin treatment

SUMMARY:
Worldwide there is an increase in antibiotic resistance which may have fatal long-term consequences. This is due to extensive use and sometimes misuse of antibiotics in the treatment of harmless infections.

The primary aim of this study is to investigate if treatment with dicloxacillin can lead to drug-drug interactions through induction of the efflux transporter P-glycoprotein (P-gp). In this study it will also be investigated whether dicloxacillin induces its own metabolism.

The hypothesis is based on a previous in vivo study showing that rifampicin induces the intestinal P-gp transporter, through activation of the pregnane X receptor (PXR). Dicloxacillin also activates the PXR receptor in vitro, which could result in an induction of P-gp in vivo.

Trial subjects will ingest dicloxacillin for 30 days and at day 10 and 28 ingest dabigatran etexilate to determine if the P-gp transporter has been induced. Plasma and urine will be drawn over 32 hours to determine the concentration of dabigatran.

Change in dicloxacillin concentration will also be measured at day 9 and 27 to establish if dicloxacillin induces its own metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* The following data must be in the normal range or only clinical insignificantly different from this: Estimated glomerular filtration rate (eGFR), alanine aminotransferase (ALAT), bilirubin, HbA1c, hemoglobin
* BMI >18.5 and < 30 kg/m2
* Bodyweight ≥ 50 kg
* Non-smoker (abstained from smoking minimum 2 weeks before the first study day and during the trial)
* Generally healthy
* Willing to give informed consent

Exclusion Criteria:

* Known sensitivity to any of the used drugs or any excipients listed in section 6.1 in the Summary of Product Characteristics (SmPC)
* Participating in any other intervention trials
* Intake of any significant prescription drugs, over-the- counter drugs, herbal drugs, or dietary supplements*. Contraindicated drugs include:

Anticoagulants, antiplatelet aggregation medicinal products, ticagrelor, clopidogrel, acetylsalicylic acid, chronic NSAIDs use, amiodarone, verapamil, systemic ketoconazole, clarithromycin, cyclosporin, itraconazole, tacrolimus, posaconazole, dronedarone, glecaprevir/pibrentasvir, quinidine, ritonavir, digoxin, selective serotonin reuptake inhibitors (SSRIs), selective serotonin norephinephrine reuptake inhibitors (SNRIs), pantoprazole, ranitidine, previous use of dicloxacillin or other P-gp or Cytochrome P450 (CYP450) inhibitors/inducers within 4 weeks prior to the start of treatment, probenecid, tetracycline, methotrexate

* Alcohol abuse or if the Danish Health Authority recommendation regarding alcohol intake has been exceeded 2 weeks before the first study day (men 14 units alcohol/week, women 7 unites alcohol/week)
* A positive pregnancy test at inclusion screening or any of the study days
* Known penicillin allergy or reactions against cephalosporins, cephamycin, 1-oxa-ß-lactamer, or carbapenems
* Women who are breastfeeding
* Diagnosis of any of the following diseases (current or previous):

Mechanical heart valve, congenital or acquired coagulation disorders, thrombocytopenia or functional platelet defects, biopsy within 4 weeks, major trauma, bacterial endocarditis, esophagitis, gastritis, gastroesophageal reflux, active meningitis, encephalitis, intracranial abscess, undergoing surgery, liver disease, history of thrombosis or diagnosed with antiphospholipid syndrome, active cancer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Change in Area under the curve (AUC) of dabigatran | Baseline and day 28
  Change in the activity of the drug transporter P-gp

SECONDARY OUTCOMES:
Change in AUC of dabigatran | Day 10 and 28
  Change in the activity of the drug transporter P-gp
Change in AUC of relevant metabolites of dabigatran etexilate | Day 10 and 28
  Change in the activity of the drug transporter P-gp
Change in Peak Plasma concentration (Cmax) of dabigatran | Day 10 and 28
  Change in the activity of the drug transporter P-gp
Change in Cmax of relevant metabolites of dabigatran etexilate | Day 10 and 28
  Change in the activity of the drug transporter P-gp
Change in Time to reach Cmax (Tmax) of dabigatran | Day 10 and 28
  Change in the activity of the drug transporter P-gp
Change in Tmax of relevant metabolites of dabigatran etexilate | Day 10 and 28
  Change in the activity of the drug transporter P-gp
Change in renal clearance (CLr) of dabigatran | Day 10 and 28
  Change in the activity of the drug transporter P-gp
Change in CLr of relevant metabolites of dabigatran etexilate | Day 10 and 28
  Change in the activity of the drug transporter P-gp
Change in Elimination half-life (T1/2) of dabigatran | Day 10 and 28
  Change in the activity of the drug transporter P-gp
Change in T1/2 of relevant metabolites of dabigatran etexilate | Day 10 and 28
  Change in the activity of the drug transporter P-gp
Change in AUC of dicloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of dicloxacillin
Change in AUC of the metabolite of dicloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of dicloxacillin
Change in Cmax of dicloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of dicloxacillin
Change in Cmax of the metabolite of dicloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of dicloxacillin
Change in Tmax of dicloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of dicloxacillin
Change in Tmax of the metabolite of dicloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of dicloxacillin
Change in CLr of dicloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of dicloxacillin
Change in CLr of the metabolite of dicloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of dicloxacillin
Change in T1/2 of dicloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of dicloxacillin
Change in T1/2 of the metabolite of dicloxacillin | Day 9 and 27
  Change in the activity of the enzyme responsible for metabolism of dicloxacillin
Change in biomarkers of drug metabolism enzymes and transporters (DMET) | 10 and 28
  Change in biomarkers for enzymes and transporters after dicloxacillin treatment
Change in exosome-derived biomarkers | 10 and 28
  Change in exosome-derived biomarkers after dicloxacillin treatment to determine activity of CYP enzymes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Denmark, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be shared due to general data protection regulation (GDPR)